CLINICAL TRIAL: NCT06063187
Title: Technology-based Fall Risk Assessments for Older Adults in Low-income Settings
Status: Completed | Type: Observational
Sponsor: University of Central Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ladda Thiamwong, Associate Professor, University of Central Florida
Other Study IDs: STUDY00002473; R03AG069799 (NIH)
Record Dates: First submitted 2023-02-07; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Fall; Physical Inactivity; Sedentary Behavior
Keywords: accidental falls; body composition; falls; fear; risk assessment; technology; wearable devices
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to examine the associations among fall risk appraisal, body composition, and physical activity in older adults in low-income settings.

The main questions it aims to answer are:

* What is the feasibility of recruitment (e.g., how many older adults need to be screened to recruit the sample?), especially during the COVID-19 pandemic, and acceptability of technologies and procedures for use among older adults in low-income settings?
* What are the the dynamic relationships between fall risk appraisal, body composition, physical activity, and behavioral changes related to fear of falling?

Participants will:

* complete questionnaires about their characteristics, socio-demographic, medical history, cognition, depressive symptoms, anxiety, and fear of falling.
* participate in static and dynamic balance tests, body composition measurement and handgrip strength test.
* wear an accelerometer for physical activity assessment for 7 consecutive days.

DETAILED DESCRIPTION:
The investigators will use a cross-sectional design to address aims. The investigators will administer the study instruments which consist of objective and subjective measures. Participants will complete questionnaires about their characteristics, socio-demographic, medical history, cognition, depressive symptoms, anxiety, and fear of falling.

Balance performance will be assessed by the BTrackS Balance System (BBS). This test consists of four, 20 seconds trials. For each trial, the participants will stand as still as possible on the BBP with hands on their hips, and eye closed. This test consists of four trials. This test will take about 5-10 minutes.

Body composition will be assessed using a bioelectrical impedance analysis (BIA): InBody S10. The BIA InBody S10 measures fat mass, muscle mass and body water levels. There are no risks, no dunking, no pinching, no discomfort associated with the use of bioelectrical impedance analysis. Test duration is 1-2 minutes.

Physical Activity (PA) will be measured by activity monitoring devices. All participants will wear the ActiGraph GT9X Link wireless activity monitor (ActiGraph LLC.), a tri-axial accelerometer, on the non-dominant wrist for 7 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years of age
* no marked cognitive impairment [Memory Impairment Screen (MIS) score ≥5]
* speak English or Spanish
* live in Kinneret Sr. Apartments or in Orlando FL.

Exclusion Criteria:

* a medical condition precluding balance test (e.g., unable to stand on the balance plate) and/or PA (e.g., shortness of breath; feeling pressure when performing PA)
* currently receiving treatment from a rehabilitation facility
* have a metal implant.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment of low-income older adults | Through study completion, an average of 2 years
  The investigators will assess the ability to recruit the participants by tracking the number of days and time spent to recruit the sample.
Acceptability of using technologies in low-income older adults | Through study completion, an average of 2 years
  The acceptability of the technologies and procedures will be examined based on an evaluation form (e.g., what the participants thought about the questionnaires and technology) and participants' recommendations.
Maladaptive fall risk appraisal | Once at baseline, an average of 5 minutes
  A condition in which there is a discrepancy between perceived fall risk (levels of fear of falling) and physiological fall risk (balance performance). Fear of falling will be assessed using the Short Fall Efficacy Scale International (short FES-I) with 7 items and balance performance will be assessed using the BTrackS Balance test. Maladaptive fall risk will be plotted on a electronic graph as the interaction between balance performance on the X-axis and fear of falling on the Y-axis.
Time spent in each physical activity intensity domain | 7 days
  Participants will wear the ActiGraph GT9X Link wireless activity monitor (ActiGraph LLC.), a tri-axial accelerometer, on the non-dominant wrist for 7 consecutive days.This device will assess the time (minutes) spent in light, moderate, and vigorous physical activity domains throughout the 7-day assessment period.
Body Composition | Once at baseline, an average of 2 minutes
  Body composition will be assessed using a direct segmental multi-frequency bioelectrical impedance analysis (BIA): InBody s10 device.
Balance Performance | Once at baseline, an average of 4 minutes
  Balance performance will be assessed using the BTrackS Balance test.
Fear of Falling | Once at baseline, an average of 10 minutes
  Fear of falling will be assessed using the Short Fall Efficacy Scale International (short FES-I) with 7 items.The minimum score possible is 7 and the maximum possible score is 28. Scores of 7-8 indicate "low concern," scores of 9-13 indicate "moderate concern," and scores of 14-28 indicate "high concern."

SECONDARY OUTCOMES:
Depression | Once at baseline, an average of 10 minutes
  Depression will be assessed using the Patient Health Questionnaire-9 (PHQ-9). The minimum possible score is 0 and the maximum possible score is 27. Scores of 0-4 indicate "minimal depression," scores of 5-9 indicate "mild depression," scores of 10-14 indicate "moderate depression," scores of 15-19 indicate "moderately severe depression," and scores of 20-27 indicate "severe depression."

CONTACTS AND LOCATIONS:
Overall Officials: Ladda Thiamwong, PhD, RN, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
The data will be made available at the end of the funding period (anticipated Fall 2023). We plan to share the de-identified datasets in both proprietary (SPSS files containing variables descriptions) and non-proprietary (.csv with accompanying .txt file containing variable descriptions) formats.

REFERENCES:
- [Background] Thiamwong L, Stout JR, Park JH, Yan X. Technology-Based Fall Risk Assessments for Older Adults in Low-Income Settings: Protocol for a Cross-sectional Study. JMIR Res Protoc. 2021 Apr 7;10(4):e27381. doi: 10.2196/27381. PMID 33825688
- [Result] Choudhury R, Park JH, Thiamwong L, Xie R, Stout JR. Objectively Measured Physical Activity Levels and Associated Factors in Older US Women During the COVID-19 Pandemic: Cross-sectional Study. JMIR Aging. 2022 Aug 22;5(3):e38172. doi: 10.2196/38172. PMID 35994346

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT06063187/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT06063187/ICF_001.pdf